CLINICAL TRIAL: NCT06036199
Title: Safety and Impact on Quality of Life of Focused Ultrasound Pallidotomy for Dyskinetic Cerebral Palsy in Pediatric and Young Adult Subjects
Brief Title: Focused Ultrasound Pallidotomy for Dyskinetic Cerebral Palsy in Pediatric and Young Adult Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Chima Oluigbo, Principal Investigator and Sponsor, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G230044
Record Dates: First submitted 2023-05-02; First posted 2023-09-13 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy, Dyskinetic; Secondary Dystonia
Keywords: High intensity focused ultrasound (HIFU); Pallidotomy
MeSH Terms: conditions — Cerebral Palsy; Dystonic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Focused Ultrasound Pallidotomy (Experimental): Pediatric and young adult patients between ages of 8 and 22 years with pharmaco-resistant secondary dystonia due to dyskinetic cerebral palsy who have Focused Ultrasound Pallidotomy
  Interventions: Device: Focused Ultrasound Pallidotomy

INTERVENTIONS:
Device: Focused Ultrasound Pallidotomy — Use of ExAblate Transcranial MR guided Focused Ultrasound as a tool for creating bilateral or unilateral lesions in the globus pallidus (GPi) in patients with treatment-refractory secondary dystonia due to dyskinetic cerebral palsy

SUMMARY:
The primary objective of the proposed study is to evaluate the safety of ExAblate Transcranial MRgFUS as a tool for creating bilateral or unilateral lesions in the globus pallidus (GPi) in patients with treatment-refractory secondary dystonia due to dyskinetic cerebral palsy

DETAILED DESCRIPTION:
The primary objective of the proposed study is to evaluate the safety of ExAblate Transcranial MRgFUS as a tool for creating bilateral or unilateral lesions in the globus pallidus (GPi) in patients with treatment-refractory secondary dystonia due to dyskinetic cerebral palsy.

The secondary is to assess the impact on Quality of Life of Focused Ultrasound Bilateral and unilateral Pallidotomy for Dyskinetic Cerebral Palsy in Pediatric and Young Adult Subjects. In addition, the impact of bilateral pallidotomy on motor development, pain perception, speech, memory, attention and cognition in these patients will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* The treating physician has chosen GPi-DBS or pallidotomy for the treatment of the secondary dystonia caused by cerebral palsy in this patient
* Patient and/or legal representative, if the patient is underaged or not capable to give consent himself, have chosen pallidotomy as treatment
* The consent to participate in the trial of the underaged patient, if he is capable to understand the study requirements, is required
* Age at enrolment 8-22 years
* Diagnosis of secondary dystonia due to cerebral palsy caused by perinatal hypoxic injury
* Anti-dystonic pharmacotherapy insufficient
* Stable anti-dystonic medication over the last 30 days
* Globus pallidus internus (pars posterior) and thalamus (motor part) intact on MRI (not older than 2 years - if possible)
* No fixed severe skeletal deformations with loss of function, which need immediate orthopaedic surgical intervention
* Sufficient compliance of the patient or the legal representative if the patient is underaged or not capable to give consent himself to take part in the study
* Informed consent to take part in the study from patient and/or legal representative if the patient is underaged or not capable to give consent himself
* Patient and/or legal representative if the patient is underaged or not capable to give consent himself, understands the study requirements and the treatment procedures and provides written informed consent before any study-specific tests or procedures are performed

Exclusion Criteria:

* Patients with known primary (e.g. DYT1) or idiopathic dystonia
* Severe axial hypotonia with total loss of head control (e.g. absence of control at "upper thoracic level" in the SATCo score) (medication effect excluded)
* Fixed hemi-dystonia
* Severe spasticity in knee- and elbow-flexors and -extensors (Modified Ashworth Scale >3)
* Fixed severe skeletal contractions with loss of function which require immediate orthopaedic surgical intervention
* Patients with other severe concurrent neurological disease (e. g. brain tumor, neurodegenerative diseases, trauma etc.)
* Condition likely to require use of MRI in the future
* Any intracranial abnormality or medical condition that would contraindicate DBS surgery
* Any findings in neuropsychological screening assessments that would contraindicate DBS surgery
* Any current drug and / or alcohol abuse
* Any history of frequent grand-mal seizures without response to anticonvulsive treatment
* Any other active implanted device (e.g. Cochlear implant, pacemaker), whether turned on or off, would be allowed provided that they do not interfere with functioning of the device.
* The presence of DBS leads due the risks of these ferromagnetic devices in the MRI environment.
* A history of neurostimulation intolerance in any area of the body.
* Currently on any anticoagulant medications that cannot be discontinued during perioperative period.
* Any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints, including any terminal illness with survival <24 months.
* Participation in another drug, device, or biologics trial concurrently or within the preceding 30 days; any other trial participation should be approved by the Principal Investigator.
* A female that is breastfeeding or of childbearing potential with a positive urine pregnancy test or - if a person is sexually active - not using sufficient contraception with a Pearl Index of less than 1% including all forms of hormonal contraception ("antibaby-pill", hormonal plaster, NuvaRing®, Implanon®, hormonal depot injections, contraceptive coil), the tubal ligature (female sterilization). Alternatively, the female of child bearing potential is sexually abstinent.
* Subjects who have contraindications to anesthesia, in the judgment of the attending anesthesiologist
* Subjects who are unwilling or unable to undergo general anesthesia
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data.
* Minimum head circumference < 49cm
* Skull Density Ratio (SDR) <0.40.

Ages: 8 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of device-related and procedure-related adverse events (AE) | 2 years
  Safety will be determined by an evaluation of the incidence and severity of device-related and procedure-related adverse events (AE) from the first treatment day visit through the 24-month post-treatment time point. All AEs will be reported and categorized as related to the device versus the ablation procedure.

SECONDARY OUTCOMES:
Burke-Fahn-Marsden-Dystonia Rating Scale movement and disability | 2 years
  Assessment of speech and swallowing. Score range: 0-30, 0 indicates complete independence, 30 indicates complete dependence.
Family Scale (FaBel) | 2 years
  Assessment of the burden for caregivers. Score range: 0-84, 0 indicates no burden, 84 indicates very severe burden.
Canadian Occupational Performance Measure (COPM) | 2 years
  Assessment of activities of daily living.
Gross Motor Function Measure (GMFM-66) | 2 years
  Assessment of physical disability. Score range: 0-3, 0 indicates no performance, 3 indicates complete performance.
Gross Motor Function Classification System (GMFCS) | 2 years
  Degree of physical impairment. Score range: 1-5, 1 indicates no limitations, 5 indicates severe limitations.
SF-36 for assessment of quality of life | 2 years
  Assessment of quality of life of subject. Score range: 0-100, 0 indicates bad health state, 100 indicates an excellent health state.
Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD) | 2 years
  Assessment of Quality of life of Caregivers and Subject. Score range: 0-100, 0 indicates a bad score, 100 indicates an excellent score.
Frenchay Dysarthria Assessment | 2 years
  Assessment of speech and swallowing. Score range:
Assessment of Cognition | 2 years
  Snijders-Oomen-Non-Verbal-Intelligence Test (SON-R)
Strengths and Difficulties Questionnaire | 2 years
  Assessment of mood and attention. Score range: 0-40, 0 indicates normal, 40 indicates abnormal.
Assessment of Attention | 2 years
  Attentional Network Test (ANT)
Assessment of cognition | 2 years
  Non-Verbal-Learning Test (NVLT)
Wong Baker Faces | 2 years
  Assessment of pain. Score range; 0-10, 0 indicates no pain, 10 indicates worst pain.
Tardieu Scale | 2 years
  Assessment of the severity of spasticity. Score range: 0-5, 0 indicates no resistance, 5 indicates no movement.
Dyskinesia Impairment Scale (DIS) | 2 years
  Assessment of the severity of chorea and dystonia. Score range: 0-576, 0 indicates no dystonia, 576 indicates very severe dystonia.
Barry Albright Dystonia Scale | 2 years
  Score range: 0-32, 0 indicates no dystonia, 32 indicates severe dystonia.

CONTACTS AND LOCATIONS:
Overall Officials: Chima Oluigbo, MD, Principal Investigator — Children's National Hospital, Washington, DC
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No